CLINICAL TRIAL: NCT03696186
Title: Selective Treatment According to Molecular Subtype of Prostate Cancer
Acronym: STAMP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAMP
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Castration-resistant Prostate Cancer; Prostate Cancer Metastatic
Keywords: Metastatic Castration-resistant Prostate Cancer; Cancer Subtype; Chemotherapy; Target Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Luminal type-1 (Active Comparator): Standard treatment
  Interventions: Drug: Luminal type-1
- Luminal type-2 (Experimental): Experimental treatment
  Interventions: Drug: Luminal type-2
- Neuroendocrine type-1 (Active Comparator): Standard treatment
  Interventions: Drug: Neuroendocrine type-1
- Neuroendocrine type-2 (Experimental): Experimental treatment
  Interventions: Drug: Neuroendocrine type-2
- Atypical type-1 (Active Comparator): Standard treatment
  Interventions: Drug: Atypical type-1
- Atypical type-2 (Experimental): Experimental treatment
  Interventions: Drug: Atypical type-2

INTERVENTIONS:
Drug: Luminal type-1 — Goserelin (3.75mg, once every 4 weeks)+Docetaxel (75 mg/m2 on day 1 every 3 weeks)+Prednisone (5 mg, twice daily)
  Arms: Luminal type-1
Drug: Luminal type-2 — Goserelin (3.75mg, once every 4 weeks)+Abiraterone (1000 mg, once daily)+Prednisone (5 mg, twice daily)
  Arms: Luminal type-2
Drug: Neuroendocrine type-1 — Goserelin (3.75mg, once every 4 weeks)+Docetaxel (75 mg/m2 on day 1 every 3 weeks)+Prednisone (5 mg, twice daily)
  Arms: Neuroendocrine type-1
Drug: Neuroendocrine type-2 — Goserelin (3.75mg, once every 4 weeks)+Carboplatin (area under the curve 5 on day 1 every 3 weeks)+Docetaxel (75 mg/m2 on day 1 every 3 weeks)+Prednisone (5 mg, twice daily)
  Arms: Neuroendocrine type-2
Drug: Atypical type-1 — Goserelin (3.75mg, once every 4 weeks)+Docetaxel (75 mg/m2 on day 1 every 3 weeks)+Prednisone (5 mg, twice daily)
  Arms: Atypical type-1
Drug: Atypical type-2 — Goserelin (3.75mg, once every 4 weeks)+Abiraterone (1000 mg, once daily)+ targeted therapy according to next Generation Sequencing (NGS)+ Prednisone (5 mg, twice daily), or Goserelin (3.75mg, once every 4 weeks)+Abiraterone+ Prednisone (5 mg, twice daily) if no druggable gene mutation detected.
  Arms: Atypical type-2

SUMMARY:
This is an open-label study that includes three substudies of random distribution. First, a sample of the primary tumor will be obtained and will be analyzed by an immunohistochemical technique to determine several markers. Depending on the expression of these markers, the patients will be characterize as group 1 (Luminal phenotype), group 2 (Neuroendocrine phenotype) or group 3 (Atypical phenotype) and a random assignment will be performed to standard or experimental treatment.

DETAILED DESCRIPTION:
Metastatic castration-resistant prostate cancer (mCRPC) is a heterogenous disease with at least 3 intrinsic subtypes including luminal, neuroendocrine, and atypical phenotypes. Different subtypes have different prognosis and treatment sensitivity. Thus, it would be more suitable to administer different therapy in different subtypes. Therefore, the investigators designed this phase 2 randomized clinical trial to explore potential effective regimens in variable subtypes of mCRPC. Patients were first classified into Luminal type, Neuroendocrine type and Atypical type by immunohistochemistry exam of FKBP5/AR-WT/AR-v7/CgA/SYN/YAP1 in core needle biopsy and then randomized to received either standard or experimental treatment.

1. Group 1 (Luminal type):

   Standard treatment: Goserelin (3.75mg, once every 4 weeks)+Docetaxel (75 mg/m2 on day 1 every 3 weeks)+Prednisone (5 mg, twice daily)

   Experimental treatment: Goserelin (3.75mg, once every 4 weeks)+Abiraterone (1000 mg, once daily)+Prednisone (5 mg, twice daily)
2. Group 2 (Neuroendocrine type):

   Standard treatment: Goserelin (3.75mg, once every 4 weeks)+Docetaxel (75 mg/m2 on day 1 every 3 weeks)+Prednisone (5 mg, twice daily)

   Experimental treatment: Goserelin (3.75mg, once every 4 weeks)+Carboplatin (area under the curve 5 on day 1 every 3 weeks)+Docetaxel (75 mg/m2 on day 1 every 3 weeks)+Prednisone (5 mg, twice daily)
3. Group 3 (Atypical type):

Standard treatment: Goserelin (3.75mg, once every 4 weeks)+Docetaxel (75 mg/m2 on day 1 every 3 weeks)+Prednisone (5 mg, twice daily)

Experimental treatment: Goserelin (3.75mg, once every 4 weeks)+Abiraterone (1000 mg, once daily)+targeted therapy according to next Generation Sequencing (NGS)+Prednisone (5 mg, twice daily); or Goserelin (3.75mg, once every 4 weeks)+Abiraterone alone+Prednisone (5 mg, twice daily) if no druggable gene mutation detected. The detailed Individual treatment see below.

The duration of chemotherapy is 6-10 cycles. Primary endpoint is the overall survival (OS) in each subtypes. Secondary endpoints include progression free survival (PFS), PSA response rate and safety. Tissue samples and blood samples will be collected at baseline and during treatment. There will be exploratory biomarkers analyses to identify predictive markers for efficacy in every subtypes.

Targeted Therapy: Participants with druggable gene mutations will receive the corresponding molecular targeted drugs.

1. Participants with epidermal growth factor receptor (EGFR) gene mutation will receive Gefitinib, which inhibits a protein called EGFR that is thought to be a key factor in the development and progression of some cancers.
2. Participants with B-type Raf kinase (BRAF) gene mutations will receive Vemurafenib, which inhibits a protein called mitogen-activated or extracellular signal-regulated protein kinase kinase (MEK) that is thought to be a key factor in the development and progression of some cancers.
3. Participants with v-akt murine thymoma viral oncogene homologue 1 (AKT1) gene mutations will receive Celecoxib, which inhibits a protein called v-akt murine thymoma viral oncogene homologue (AKT) that is thought to be a key factor in the development and progression of some cancers.
4. Participants who have erythroblastic leukemia viral oncogene homolog 2 (ERBB2) gene mutation will receive Lapatinib, which inhibits some proteins that are thought to be key factors in the development and progression of some cancers.
5. Participants with PDGFRA/PDGFRB gene mutations will receive Sunitinib, which inhibits some proteins that are thought to be key factors in the development and progression of some cancers.
6. Participants with PIK3CA gene mutations will receive Everolimus, which inhibits a protein called AKT that is thought to be a key factor in the development and progression of some cancers.
7. Participants with DNA-repair gene defects will receive Olaparib, which inhibits poly ADP ribose polymerase (PARP).

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have given consent form;
2. Patients with a confirmed diagnosis of mCRPC according to EAU 2018 guideline;
3. Serum testosterone must reach castration level: <50 ng per deciliter;
4. Participants with life expectancy of at least 6 months based on the Investigator's clinical judgment.

Exclusion Criteria:

1. Participants who are allergic to contrast medium;
2. Patients were excluded if they planned to receive additional concurrent anticancer therapies;
3. Patients doesn't sign an informed consent form.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 40 months
  OS was defined as the duration from the initiation of treatment to death of any cause

SECONDARY OUTCOMES:
PSA-Progression free survival (pPFS) | Up to 40 months
  PSA progression was defined as an increase in the PSA level of 25% or more above the nadir (and by≥2 ng/ml), with confirmation of 4 or more weeks later
Radiographic progression free survival (rPFS) | Up to 40 months
  rPFS was defined 1) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria; or 2) as at least two new lesions on first post-treatment bone scan, with at least two additional lesions on the next bone scan
PSA response rate | Up to 40 months
  PSA response is defined as ≥ 50% decline in PSA level from baseline, maintained for≥ 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, China